CLINICAL TRIAL: NCT05931367
Title: A Phase 3 Study to Investigate the Efficacy and Safety of LY3437943 Once Weekly in Participants Who Have Obesity or Overweight and Osteoarthritis of the Knee: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: A Study of Retatrutide (LY3437943) Once Weekly in Participants Who Have Obesity or Overweight and Osteoarthritis of the Knee
Acronym: TRIUMPH-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18583; J1I-MC-GZBN (Other: Eli Lilly and Company); 2023-503660-17-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-06-27; First posted 2023-07-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obesity; Overweight; Osteo Arthritis Knee
MeSH Terms: conditions — Obesity; Overweight | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Retatrutide Dose 1 (Experimental): Participants will receive retatrutide subcutaneously (SC).
  Interventions: Drug: Retatrutide
- Retatrutide Dose 2 (Experimental): Participants will receive retatrutide SC.
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide Dose 1; Retatrutide Dose 2
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of retatrutide once-weekly in participants who have obesity or are overweight and have osteoarthritis (OA) of the knee. The study will lasts about 77 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) ≥27 kilogram/kg/m² at screening.
* Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight.
* Have index knee pain for >12 weeks prior to screening, and presence of index knee pain for >15 days over the previous month.
* Have knee X-ray with moderate radiographic changes (Kellgren-Lawrence Grade 2 or 3) per central reading at screening.
* Currently meets American College of Rheumatology (ACR) Criteria (clinical and radiological) for OA.

Exclusion Criteria:

* Have had steroid joint injections within 90 days of screening.
* Have had other joint injections and procedures within 6 months of screening.
* Have joint disease other than osteoarthritis.
* Have a self-reported or documented change in body weight >5 kg (11 pounds) within 90 days prior to screening.
* Have been taking weight loss drugs, including over-the-counter medications, within 90 days prior to screening.
* Have a prior or planned surgical treatment for obesity.
* Have diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score | Baseline, Week 68
Percent Change from Baseline in Body Weight | Baseline, Week 68

SECONDARY OUTCOMES:
Change from Baseline in the WOMAC Physical Function Subscale Score | Baseline, Week 68
Change from Baseline in Waist Circumference | Baseline, Week 68
Percent Change from Baseline in Total Cholesterol | Baseline, Week 68
Percent Change from Baseline in Triglycerides | Baseline, Week 68
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 68
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 68
Change from Baseline in Diastolic Blood Pressure (DBP) | Baseline, Week 68
Percent Change from Baseline in Fasting Insulin | Baseline, Week 68
Change from Baseline in Short Form 36-Version 2 (SF-36v2) Acute Form Physical Functioning Domain Score | Baseline, Week 68
Change from Baseline in Average Pain Intensity Numeric Rating Score (API-NRS) Score | Baseline, Week 68
Change from Baseline in Worst Pain Intensity Numeric Rating Score (WPI-NRS) Score | Baseline, Week 68

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (13):
  - Arizona Research Center, Phoenix, Arizona
  - Artemis Institute for Clinical Research, San Diego, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Suncoast Research Group, Miami, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Northwestern University, Chicago, Illinois
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Clinvest Research LLC, Springfield, Missouri
  - Mercy Family Clinic, Dallas, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Australia (8):
  - Paratus Clinical Research Canberra, Bruce, Australian Capital Territory
  - Paratus Clinical Research Western Sydney, Blacktown, New South Wales
  - Emeritus Research, Botany, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Core Research Group, Brisbane, Queensland
  - CDH Research Institute, Maroochydore, Queensland
  - Emeritus Research, Camberwell, Victoria
  - Barwon Health, Geelong, Victoria
- Canada (10):
  - C-health Research, Calgary, Alberta
  - Eastern Health - General Hospital, St. John's, Newfoundland and Labrador
  - Viable Clinical Research, Bridgewater, Nova Scotia
  - Wharton Medical Clinic, Hamilton, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Viable Clinical Research, Scarborough Village, Ontario
  - Stouffville Medical Research Institute Inc., Stouffville, Ontario
  - Canadian Phase Onward, Toronto, Ontario
  - Alpha Recherche Clinique, Québec
  - ALPHA Recherche Clinique, Québec
- Mexico (7):
  - Consultorio Médico, Guadalajara, Jalisco
  - IMED Internal Medicine Clin Trials, Monterrey, Nuevo León
  - Clínica García Flores SC, Monterrey, Nuevo León
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza, Nuevo León
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero, Tamaulipas
  - Kohler and Milstein Research S.A. de C.V., Mérida, Yucatán
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
- Spain (8):
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval"), Ferrol, A Coruña
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Quirón Málaga, Málaga, Andalusia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital General Universitario de Valencia, Valencia, Valenciana
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
- United Kingdom (3):
  - Leicester General Hospital, Leicester, Leicestershire
  - Panthera Biopartners - North London, Enfield, London
  - Panthera Biopartners - Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) Once Weekly in Participants Who Have Obesity or Overweight and Osteoarthritis of the Knee (TRIUMPH-4) — https://trials.lilly.com/en-US/trial/408355